CLINICAL TRIAL: NCT05899933
Title: Implantoplasty Versus Implant Decontamination With Erythritol Air-abrasive Device During Surgical Therapy of Peri-implantitis. Clinical, Radiographic and Microbiological Evaluation. A Randomized Controlled Clinical Study
Brief Title: Comparison of the Effectiveness of Two Different Surgical Therapeutic Protocols of Peri-implantitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Yiorgos A. Bobetsis, Assistant Professor, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PERIO1
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Peri-Implantitis; Peri-Implant Health
Keywords: Peri-Implantitis; Surgical therapy; Implantoplasty; Air-abrasive device; Erythritol powder; Peri-Implant microbiota
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: The experimental protocol is designed as a double-blind, randomized clinical trial with a 12-month duration and a parallel design
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Implantoplasty group (Experimental): 6 weeks after completion of non-surgical peri-implant therapy, participants with peri-implant probing pocket depth ≥ 5mm and presence of bleeding on probing and/or suppuration will receive resective surgical treatment. Implantoplasty will be applied as an implant surface modification method.
  Interventions: Procedure: Non-surgical peri-implant therapy; Procedure: Implantoplasty; Procedure: Prophylaxis
- Erythritol Air-abrasive device group (Experimental): 6 weeks after completion of non-surgical peri-implant therapy, participants with peri-implant probing pocket depth ≥ 5mm and presence of bleeding on probing and/or suppuration will receive resective surgical treatment. Implant surface decontamination with an air-abrasive device with erythritol powder will be applied.
  Interventions: Procedure: Non-surgical peri-implant therapy; Procedure: Erythritol Air-abrasive device; Procedure: Prophylaxis
- Control group (Other): Participants with healthy implants will be the comparator group for the microbiological analysis.
  Interventions: Procedure: Prophylaxis

INTERVENTIONS:
Procedure: Non-surgical peri-implant therapy — 2 weeks after baseline examination, non surgical therapy will be applied in implants diagnosed with peri-implantitis prior to enrollment in surgical therapy.
  Firstly, participants will be instructed in oral hygiene. Professional supragingival and subgingival debridement of implants/ teeth, including the selected for the study implants, will be performed. Local anesthesia will be performed, when needed. Targeted implants will be treated with PEEK-coating ultrasonic tips (Instrument PI; EMS), titanium curettes (IMPM11/12T, IMPM13/14T; Hu-Friedy), rubber cup and polishing paste. Possible adjustments to implant-borne prostheses will be considered, whenever possible. Re-evaluation of non-surgical therapy will be performed after 6 weeks.
  At the 6-week reevaluation, participants with peri-implant probing pocket depth ≥5 mm and bleeding on probing and/or suppuration in patients with full mouth plaque score ≤20% will proceed to surgical therapy.
  Arms: Erythritol Air-abrasive device group; Implantoplasty group
Procedure: Implantoplasty — Screw-retained supraconstructions and, when possible, cement-retained restorations will be removed.
  Following local anesthesia, intrasulcular incisions will be performed and full-thickness flaps will be elevated on the buccal and lingual aspects of affected implants. Granulation tissue will be removed, and titanium-coated curettes (IMPM11/12T, IMPM13/14T; Hu-Friedy) and NiTi brushes (NEGRIN IN DENTAL) will be applied to remove hard deposits on implants. Osseous recontouring will be performed when indicated followed by irrigations with saline. Implantoplasty will be applied using tungsten carbide burs of various shapes and sizes (Peri-implantitis Kit; Meisinger) followed by irrigations with saline. Flaps will be readjusted and closed with sutures in order to allow a non-submerged healing. Supraconstructions will be reconnected after the surgery.
  Arms: Implantoplasty group
Procedure: Erythritol Air-abrasive device — Screw-retained supraconstructions and, when possible, cement-retained restorations will be removed.
  Following local anesthesia, intrasulcular incisions will be performed and full-thickness flaps will be elevated on the buccal and lingual aspects of affected implants. Granulation tissue will be removed, and titanium-coated curettes (IMPM11/12T, IMPM13/14T; Hu-Friedy), and NiTi brushes (NEGRIN IN DENTAL) will be applied to remove hard deposits on implants. Osseous recontouring will be performed when indicated followed by irrigations with saline. Implant surface decontamination with an air-abrasive device (AIRFLOW® MAX, AIRFLOW® Prophylaxis Master; EMS) with erythritol powder (AIRFLOW® Plus Powder; EMS) will be applied followed by irrigations with saline. Flaps will be readjusted and closed with sutures in order to allow a non-submerged healing. Supraconstructions will be reconnected after the surgery.
  Arms: Erythritol Air-abrasive device group
Procedure: Prophylaxis — Supramucosal biofilm removal of implants/ teeth will be performed at, 3, 6, 9 and 12 months after surgical therapy for the Implantoplasty group and the Erythritol Air-abrasive device group and at 2 weeks, 3, 6, 9 and 12 months after baseline examination for the control group. Targeted implants will be treated with an air-abrasive device (AIRFLOW® MAX, AIRFLOW® Prophylaxis Master; EMS) with erythritol powder (AIRFLOW® Plus Powder; EMS). During these appointments, patients will be re-motivated and re-instructed to oral-hygiene measures.

SUMMARY:
The purpose of the present study is to compare the 1-year clinical, radiographic and microbiological outcomes and patients' satisfaction following surgical treatment of peri-implantitis after applying two different surface modification methods. Secondarily, analysis and comparison of the microbiological results of implants diagnosed and treated for peri-implantitis with healthy implants will be performed.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* Participants ≥ 18 years and ≤ 80 years of age
* Non-smokers based on the patients' self-reported smoking status, defined as patients who had never smoked or had quit smoking at least 2 years ago
* Implants in function for more than 1 year after suprastructure connection

Inclusion Criteria for implants diagnosed with Peri-Implantitis:

* Presence of at least one implant diagnosed with peri-implantitis defined as presence of bleeding on probing and/or suppuration, probing pocket depth ≥6 mm and ≥3 mm of detectable bone loss after initial re-modelling
* Absence of implant mobility

  * in participants with more than one implant, the implant with the worst clinical condition will be studied.

Inclusion Criteria for implants diagnosed with Peri-Implant Health:

* Absence of peri-implant signs of inflammation (redness, swelling)
* Lack of bleeding on probing
* Absence of bone loss beyond crestal bone level changes resulting from initial remodeling, which should not be ≥2 mm

Exclusion Criteria:

* Smokers
* Uncontrolled diabetes mellitus (HBA1c >7)
* Treatment with bisphosphonates
* Needing antibiotic prophylaxis
* Currently pregnant or breast-feeding women
* History of systemic administration of antibiotic treatment during the preceding 3 months
* Systemic conditions that contraindicate treatment
* Use of medications known to induce gingival hyperplasia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Treatment success as described by the composite outcome of probing pocket depth (PPD) ≤5 mm, absence of bleeding on probing (BoP) and/or suppuration and bone loss ≤0.5 mm between week 2 and 12 months post-surgery, at 12-month examination post-surgery | 12 months post-surgery
  The percentage of treatment success will be calculated from the total amount of treated implants.
  * PPD will be measured in mm as the distance from the mucosal peri-implant margin to the bottom of the probeable peri-implant pocket with a manual periodontal probe to the closest millimeter at the mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual site of the targeted implants.
  * BoP will be assessed dichotomously (1=presence, 0=absence) within 30 seconds after probing at the mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual site of the targeted implants.
  * Mean change in mm in mean marginal bone level (mesial and distal) will be assessed using an image-processing software.
  Standardized intra-oral radiographs will be obtained at each time point using a reproducible technique.
  Marginal bone level will be calculated as the distance from the implant shoulder to the most coronal bone-to-implant contact.
Mean total colony forming units (CFU) counts of the bacterial species under study in targeted implants with peri-implantitis from Baseline to Week 6 after non-surgical therapy | Baseline, Week 6 after non-surgical therapy
  Mean total CFU counts from Baseline to Week 6 after non-surgical therapy will be assessed at each experimental group.
  Mean total CFU counts will result from microbiological analysis of subgingival samples by quantitative PCR (qPCR).
  Subgingival samples will be obtained with three sterile paper points from the deepest pocket of targeted implants at Baseline and at Week 6 after completion of non-surgical therapy.
  Detection and quantification of bacterial DNA of Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola, Prevotella intermedia, Fusobacterium nucleatum and Campylobacter rectus will be performed.
Mean total colony forming units (CFU) counts of the bacterial species under study in targeted implants with peri-implantitis from Baseline to 12 months after surgical therapy | Baseline, 3 months post-surgery, 6 months post-surgery, 12 months post-surgery
  Mean total CFU counts from Baseline to 12 months after surgical therapy will be assessed at each experimental group.
  Mean total CFU counts will result from microbiological analysis of subgingival samples by quantitative PCR (qPCR).
  Subgingival samples will be obtained with three sterile paper points from the deepest pocket of targeted implants at Baseline, 3 months post-surgery, 6 months post-surgery and 12 months post-surgery.
  Detection and quantification of bacterial DNA of Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola, Prevotella intermedia, Fusobacterium nucleatum and Campylobacter rectus will be performed.
Mean total colony forming units (CFU) counts of the bacterial species under study in targeted implants of the control group from Baseline to 12 months follow-up visit | Baseline, 3 months follow-up visit, 6 months follow-up visit, 12 months follow-up visit
  Mean total CFU counts from Baseline to 12 months after Baseline examination will be assessed.
  Mean total CFU counts will result from microbiological analysis of subgingival samples by quantitative PCR (qPCR).
  Subgingival samples will be obtained with three sterile paper points from the implant site with the easiest access for sampling at Baseline, 3 months follow-up visit, 6 months follow-up visit, 12 months follow-up visit.
  Detection and quantification of bacterial DNA of Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola, Prevotella intermedia, Fusobacterium nucleatum and Campylobacter rectus will be performed.

SECONDARY OUTCOMES:
Mean peri-implant probing pocket depth from Baseline to Week 6 after non-surgical therapy | Baseline, Week 6 after non-surgical therapy
  Mean peri-implant probing pocket depth (PPD) will be assessed at Baseline examination and Week 6 after non-surgical therapy.
  At each examination, PPD will be recorded at six sites per targeted implant. PPD will be measured in mm as the distance from the mucosal peri-implant margin to the bottom of the probeable peri-implant pocket with a manual periodontal probe to the closest millimeter at the mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual site of the studied implant.
Mean peri-implant probing pocket depth from Baseline to 12 months after surgical therapy | Baseline, 3 months post-surgery, 6 months post-surgery, 12 months post-surgery
  Mean peri-implant probing pocket depth (PPD) will be assessed at Baseline examination and 12 months after surgical therapy.
  At each examination, PPD will be recorded at six sites per targeted implant. PPD will be measured in mm as the distance from the mucosal peri-implant margin to the bottom of the probeable peri-implant pocket with a manual periodontal probe to the closest millimeter at the mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual site of the studied implant.
Mean change from Baseline in peri-implant probing pocket depth at Week 6 after non-surgical therapy | Baseline, Week 6 after non-surgical therapy
  Mean change in mm in peri-implant probing pocket depth (PPD) will be assessed between Baseline examination and Week 6 after non-surgical therapy.
  At each examination, PPD will be recorded at six sites per targeted implant. PPD will be measured in mm as the distance from the mucosal peri-implant margin to the bottom of the probeable peri-implant pocket with a manual periodontal probe to the closest millimeter at the mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual site of the studied implant.
Mean change from Baseline in peri-implant probing pocket depth to 12 months after surgical therapy | Baseline, 3 months post-surgery, 6 months post-surgery, 12 months post-surgery
  Mean change in mm in peri-implant probing pocket depth (PPD) will be assessed between Baseline and 12 months after completion of surgical therapy.
  PPD will be recorded at six sites per targeted implant. PPD will be measured in mm as the distance from the mucosal peri-implant margin to the bottom of the probeable peri-implant pocket with a manual periodontal probe to the closest millimeter at the mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual site of the studied implant.
Percentage of sites with bleeding on probing from Baseline to Week 6 after non-surgical therapy | Baseline, Week 6 after non-surgical therapy
  Bleeding on probing will be assessed dichotomously as present (1 for bleeding presence) or absent (0 for bleeding absence) within 30 seconds after probing.
  BoP will be recorded at 6 sites per targeted implants (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual)
Percentage of sites with bleeding on probing from Baseline to 12 months after surgical therapy | Baseline, 3 months post-surgery, 6 months post-surgery, 12 months post-surgery
  Bleeding on probing will be assessed dichotomously as present (1 for bleeding presence) or absent (0 for bleeding absence) within 30 seconds after probing.
  BoP will be recorded at 6 sites per targeted implants (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual)
Change from Baseline in bleeding index score at Week 6 after completion of non-surgical therapy | Baseline, Week 6 after non-surgical therapy
  Change in percentage of sites with bleeding index score (BI) from 0 to 3 will be recorded between Baseline and Week 6 after completion of non-surgical therapy.
  BI will be recorded at 6 sites per targeted implants (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual) within 30 seconds after probing.
  Bleeding will be graded as: 0= no bleeding, 1= dot of bleeding, 2= line of bleeding, 3= profuse bleeding.
Change from Baseline in bleeding index score to 12 months after surgical therapy | Baseline, 3 months post-surgery, 6 months post-surgery, 12 months post-surgery
  Change in percentage of sites with bleeding index score (BI) from 0 to 3 will be recorded between Baseline and 12 months after completion of surgical therapy.
  BI will be recorded at 6 sites per targeted implants (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual) within 30 seconds after probing.
  Bleeding will be graded as: 0= no bleeding, 1= dot of bleeding, 2= line of bleeding, 3= profuse bleeding
Percentage of sites with suppuration on probing from Baseline to Week 6 after non-surgical therapy | Baseline, Week 6 after non-surgical therapy
  Suppuration on probing (SoP) will be assessed dichotomously as present (1 for suppuration presence) or absent (0 for suppuration absence) within 30 seconds after probing.
  SoP will be recorded at 6 sites per targeted implants (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual)
Percentage of sites with suppuration on probing from Baseline to 12 months after surgical therapy | Baseline, 3 months post-surgery, 6 months post-surgery, 12 months post-surgery
  Suppuration on probing (SoP) will be assessed dichotomously as present (1 for suppuration presence) or absent (0 for suppuration absence) within 30 seconds after probing.
  SoP will be recorded at 6 sites per targeted implants (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual)
Mean change in marginal bone level at the implant site between Week 2 after surgery and 12 months after surgery measured in intraoral radiographs | Week 2 post-surgery, 12 months post-surgery
  Mean change in mm between week 2 and 12 months post-surgery in mean marginal bone level (mesial and distal) will be assessed using an image-processing software.
  Standardized intra-oral radiographs will be obtained at Week 2 post-surgery and at 12 months post-surgery examination, using a reproducible technique with an occlusal bite index with acrylic resin mounted on a film holder.
  Marginal bone level will be calculated as the distance from the implant shoulder to the most coronal bone-to-implant contact, measured at the mesial and distal aspects of the studied implants at each time-point.
Mean peri-implant clinical attachment level from Baseline to Week 6 after non-surgical therapy | Baseline, Week 6 after non-surgical therapy
  Mean change in mm in peri-implant clinical attachment level (CAL) will be assessed at Baseline examination and Week 6 after non-surgical therapy.
  CAL will be recorded at six sites per targeted implant. CAL will be measured in mm as the distance from the most apical portion of the crown or the prosthetic connection platform for removable implant-supported restorations to the bottom of the probeable peri-implant pocket with a manual periodontal probe to the closest millimeter at the mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual site of the studied implant.
Mean peri-implant clinical attachment level from Baseline to 12 months after surgical therapy | Baseline, 3 months post-surgery, 6 months post-surgery, 12 months post-surgery
  Mean change in mm in peri-implant clinical attachment level (CAL) will be assessed at Baseline examination and Week 6 after non-surgical therapy.
  CAL will be recorded at six sites per targeted implant. CAL will be measured in mm as the distance from the most apical portion of the crown or the prosthetic connection platform for removable implant-supported restorations to the bottom of the probeable peri-implant pocket with a manual periodontal probe to the closest millimeter at the mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual site of the studied implant.
Mean change from Baseline in peri-implant clinical attachment level to Week 6 after surgical therapy | Baseline, Week 6 after non-surgical therapy
  Mean change in mm in peri-implant clinical attachment level (CAL) will be assessed from Baseline examination to Week 6 after completion of surgical therapy.
  CAL will be recorded at six sites per targeted implant. CAL will be measured in mm as the distance from the most apical portion of the crown or the prosthetic connection platform for removable implant-supported restorations to the bottom of the probeable peri-implant pocket with a manual periodontal probe to the closest millimeter at the mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual site of the studied implant.
Mean change from Baseline in peri-implant clinical attachment level to 12 months after surgical therapy | Baseline, 3 months post-surgery, 6 months post-surgery, 12 months post-surgery
  Mean change in mm in peri-implant clinical attachment level (CAL) will be assessed from Baseline examination to 12 months after completion of surgical therapy.
  CAL will be recorded at six sites per targeted implant. CAL will be measured in mm as the distance from the most apical portion of the crown or the prosthetic connection platform for removable implant-supported restorations to the bottom of the probeable peri-implant pocket with a manual periodontal probe to the closest millimeter at the mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual site of the studied implant.
Mean peri-implant recession from Baseline to Week 6 after non-surgical therapy | Baseline, Week 6 after non-surgical therapy
  Mean peri-implant recession (REC) in mm will be assessed at Baseline examination and Week 6 after non-surgical therapy.
  REC will be recorded at six sites per targeted implant. REC will be measured in mm as the distance from the free marginal mucosa to the most apical portion of the crown or the prosthetic connection platform for removable implant- supported restorations with a manual periodontal probe to the closest millimeter at the mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual site of the studied implant.
Mean peri-implant recession from Baseline to 12 months after surgical therapy | Baseline, 3 months post-surgery, 6 months post-surgery, 12 months post-surgery
  Mean peri-implant recession (REC) will be assessed in mm from Baseline examination to 12 months after surgical therapy.
  REC will be recorded at six sites per targeted implant. REC will be measured in mm as the distance from the free marginal mucosa to the most apical portion of the crown or the prosthetic connection platform for removable implant- supported restorations with a manual periodontal probe to the closest millimeter at the mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual site of the studied implant.
Mean change from Baseline in peri-implant recession at Week 6 after non-surgical therapy | Baseline, Week 6 after non-surgical therapy
  Mean change in mm in peri-implant recession (REC) will be assessed between Baseline examination and Week 6 after non-surgical therapy.
  REC will be recorded at six sites per targeted implant. REC will be measured in mm as the distance from the free marginal mucosa to the most apical portion of the crown or the prosthetic connection platform for removable implant- supported restorations with a manual periodontal probe to the closest millimeter at the mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual site of the studied implant.
Mean change from Baseline in peri-implant recession to 12 months after surgical therapy | Baseline, 3 months post-surgery, 6 months post-surgery, 12 months post-surgery
  Mean change in mm in peri-implant recession (REC) will be assessed from Baseline examination to 12 months after completion of surgical therapy.
  REC will be recorded at six sites per targeted implant. REC will be measured in mm as the distance from the free marginal mucosa to the most apical portion of the crown or the prosthetic connection platform for removable implant- supported restorations with a manual periodontal probe to the closest millimeter at the mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual site of the studied implant.
Mean local plaque score from Baseline to Week 6 after non-surgical therapy | Baseline, Week 6 after non-surgical therapy
  Mean number of sites with plaque presence at targeted implants will be assessed between Baseline examination and Week 6 after non-surgical therapy.
  Local plaque score (LPS) will be calculated by assigning a binary score at each implant surface (1 for plaque presence, 0 for plaque absence) Presence or absence of plaque will be recorded at four sites per targeted implant (mesial, buccal, distal, lingual)
Mean local plaque score from Baseline to 12 months after surgical therapy | Baseline, 3 months post-surgery, 6 months post-surgery, 12 months post-surgery
  Mean number of sites with plaque presence at targeted implants will be assessed from Baseline to 12 months after completion of surgical therapy.
  Local plaque score (LPS) will be calculated by assigning a binary score at each surface ( 1 for plaque presence, 0 for plaque absence) and calculating the percentage of total tooth/ implant surfaces with plaque presence.
  Presence or absence of plaque will be recorded at 4sites per tooth/ implant (mesial, buccal, distal, lingual)
Full mouth plaque score from Baseline to Week 6 after non-surgical therapy | Baseline, Week 6 after non-surgical therapy
  Percentage of full mouth plaque score (FMPS) presence from Baseline to Week 6 after completion of non-surgical therapy.
  FMPS will be calculated by assigning a binary score at each surface ( 1 for plaque presence, 0 for plaque absence) and calculating the percentage of total tooth/ implant surfaces with plaque presence.
  Presence or absence of plaque will be recorded at four sites per tooth/ implant (mesial, buccal, distal, lingual)
Full mouth plaque score from Baseline to 12 months after surgical therapy | Baseline, 3 months post-surgery, 6 months post-surgery, 12 months post-surgery
  Percentage of full mouth plaque score (FMPS) presence from Baseline to 12 months after completion of surgical therapy.
  FMPS will be calculated by assigning a binary score at each surface ( 1 for plaque presence, 0 for plaque absence) and calculating the percentage of total tooth/ implant surfaces with plaque presence.
  Presence or absence of plaque will be recorded at 4sites per tooth/ implant (mesial, buccal, distal, lingual)
Full mouth bleeding score from Baseline to Week 6 after non-surgical therapy | Baseline, Week 6 after non-surgical therapy
  Percentage of full mouth bleeding score (FMBS) presence from Baseline to Week 6 after completion of non-surgical therapy.
  FMBS will be calculated by assigning a binary score at each surface ( 1 for bleeding presence, 0 for bleeding absence) within 30 seconds after probing and calculating the percentage of total tooth/ implant surfaces that bled upon probing.
  Presence or absence of bleeding will be recorded at six sites per tooth/ implant (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual)
Full mouth bleeding score from Baseline to 12 months after surgical therapy | Baseline, 3 months post-surgery, 6 months post-surgery, 12 months post-surgery
  Percentage of full mouth bleeding score (FMBS) presence from Baseline to 12 months after completion of surgical therapy.
  FMBS will be calculated by assigning a binary score at each surface ( 1 for bleeding presence, 0 for bleeding absence) within 30 seconds after probing and calculating the percentage of total tooth/ implant surfaces that bled upon probing.
  Presence or absence of bleeding will be recorded at 6 sites per tooth/ implant (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual)
Evaluation of participants' pain on the visual analogue scale (VAS, 10cm) at Week 2 post-surgery | Week 2 post-surgery
  Participants will complete a questionnaire at Week 2 post-surgery in order to assess the intensity of post-surgical pain using a visual analogue scale (VAS, 10cm). The following question will be asked:
  -From 0-10, rate the intensity of pain after surgery in the treated areas. (0 represents "no pain" and 10 represents "unbearable pain").
Evaluation of participants' pain on the visual analogue scale (VAS, 10cm) at 12 months post-surgery | 12 months post-surgery
  Participants will complete a questionnaire at 12 months post-surgery in order to assess the intensity of pain at the treated sites at 12 months after surgery using a visual analogue scale (VAS, 10cm). The following question will be asked:
  From 0-10, rate the intensity of pain after surgery in the treated areas. (0 represents "no pain" and 10 represents "unbearable pain").
Evaluation of participants' pain during toothbrushing on the visual analogue scale (VAS, 10cm) at 12 months post-surgery | 12 months post-surgery
  Participants will complete a questionnaire at 12 months post-surgery in order to assess the intensity of pain during toothbrushing at the treated sites at 12 months after surgery using a visual analogue scale (VAS, 10cm). The following question will be asked:
  From 0-10, rate the intensity of pain after surgery in the treated areas. (0 represents "no pain" and 10 represents "unbearable pain").
Evaluation of participants' swelling on the visual analogue scale (VAS) at Week 2 post-surgery | Week 2 post-surgery
  Participants will complete a questionnaire at Week 2 post-surgery in order to assess the intensity of post-surgical swelling using a visual analogue scale (VAS, 10cm). The following question will be asked:
  -From 0-10 rate the amount of post-surgery swelling in the treated areas. (0 represents "no swelling" and 10 "maximum swelling").
Evaluation of participants' bleeding tendency when applying oral hygiene on the visual analogue scale (VAS, 10cm) at 12 months post-surgery | 12 months post-surgery
  Participants will complete a questionnaire at 12 months post-surgery in order to assess the intensity of bleeding during toothbrushing or interdental cleaning at the treated sites at 12 months after surgery using a visual analogue scale (VAS, 10cm). The following question will be asked:
  assess the presence and intensity of pain during toothbrushing at the treated sites at 12 months after surgery using a visual analogue scale (VAS, 10cm). The following question will be asked:
  -From 0-10 rate the amount of bleeding when applying oral hygiene to the areas you treated. (0 represents "no bleeding" and 10 "maximum bleeding").
Number of days of analgesic consumption at Week 2 post-surgery | Week 2 post-surgery
  Participants will complete a questionnaire at Week 2 post-surgery in order to record the number of days analgesics were needed .
Evaluation of patients' satisfaction on the visual analogue scale (VAS) at Week 2 post-surgery | Week 2 post-surgery
  Participants will complete a questionnaire at Week 2 post-surgery in order to assess satisfaction with the treatment provided using a visual analogue scale (VAS, 10cm). The followed questions will be asked:
  -If necessary, would you do this treatment again? (0 represents aversion to repeating the treatment and 10 that you would repeat it comfortably).
Evaluation of patients' willingness to recommend the treatment on the visual analogue scale (VAS) at Week 2 post-surgery | Week 2 post-surgery
  Participants will complete a questionnaire at Week 2 post-surgery in order to assess satisfaction with the treatment provided using a visual analogue scale (VAS, 10cm). The followed questions will be asked:
  -Would you recommend the treatment to a relative or friend? (0 represents that you would not recommend it under any circumstances and 10 that you would absolutely recommend it, if necessary).
Evaluation of patients' satisfaction on the visual analogue scale (VAS) at 12 months post-surgery | 12 months post-surgery
  Participants will complete a questionnaire at 12 months post-surgery in order to assess satisfaction with the treatment provided using a visual analogue scale (VAS, 10cm). The followed questions will be asked:
  -Are you satisfied with the treatment you received? (0 represents "not at all satisfied" and 10 "completely satisfied").
Evaluation of patients' willingness to recommend the treatment on the visual analogue scale (VAS) at 12 months post-surgery | 12 months post-surgery
  Participants will complete a questionnaire at 12 months post-surgery in order to assess satisfaction with the treatment provided using a visual analogue scale (VAS, 10cm). The followed questions will be asked:
  -Would you recommend the treatment to a relative or friend? (0 represents that you would not recommend it under any circumstances and 10 that you would absolutely recommend it, if necessary).

CONTACTS AND LOCATIONS:
Overall Officials: Phoebus N. Madianos, Study Chair — National and Kapodistrian University of Athens
Locations (1):
- Department of Periodontology, School of Dentistry, National and Kapodistrian University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes
The data that supports the findings of this study will be available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests will be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered.
Access Criteria: Access to trial individual participant data (IPD) can be requested by qualified investigators whose proposed research has received Institutional Review Board (IRB) approval. Data will be available via a data repository following execution of data use agreement.

REFERENCES:
- [Background] Carcuac O, Derks J, Charalampakis G, Abrahamsson I, Wennstrom J, Berglundh T. Adjunctive Systemic and Local Antimicrobial Therapy in the Surgical Treatment of Peri-implantitis: A Randomized Controlled Clinical Trial. J Dent Res. 2016 Jan;95(1):50-7. doi: 10.1177/0022034515601961. Epub 2015 Aug 18. PMID 26285807
- [Background] Casado PL, Otazu IB, Balduino A, de Mello W, Barboza EP, Duarte ME. Identification of periodontal pathogens in healthy periimplant sites. Implant Dent. 2011 Jun;20(3):226-35. doi: 10.1097/ID.0b013e3182199348. PMID 21613949
- [Background] Charalampakis G, Belibasakis GN. Microbiome of peri-implant infections: lessons from conventional, molecular and metagenomic analyses. Virulence. 2015;6(3):183-7. doi: 10.4161/21505594.2014.980661. Epub 2015 Feb 5. PMID 25654499
- [Background] Charalampakis G, Rabe P, Leonhardt A, Dahlen G. A follow-up study of peri-implantitis cases after treatment. J Clin Periodontol. 2011 Sep;38(9):864-71. doi: 10.1111/j.1600-051X.2011.01759.x. Epub 2011 Jul 19. PMID 21770994
- [Background] Dabdoub SM, Tsigarida AA, Kumar PS. Patient-specific analysis of periodontal and peri-implant microbiomes. J Dent Res. 2013 Dec;92(12 Suppl):168S-75S. doi: 10.1177/0022034513504950. Epub 2013 Oct 24. PMID 24158341
- [Background] Heitz-Mayfield LJ, Mombelli A. The therapy of peri-implantitis: a systematic review. Int J Oral Maxillofac Implants. 2014;29 Suppl:325-45. doi: 10.11607/jomi.2014suppl.g5.3. PMID 24660207
- [Background] Lasserre JF, Brecx MC, Toma S. Implantoplasty Versus Glycine Air Abrasion for the Surgical Treatment of Peri-implantitis: A Randomized Clinical Trial. Int J Oral Maxillofac Implants. 2020 Jan/Feb;35(35):197-206. doi: 10.11607/jomi.6677. PMID 31923303
- [Background] Maximo MB, de Mendonca AC, Renata Santos V, Figueiredo LC, Feres M, Duarte PM. Short-term clinical and microbiological evaluations of peri-implant diseases before and after mechanical anti-infective therapies. Clin Oral Implants Res. 2009 Jan;20(1):99-108. doi: 10.1111/j.1600-0501.2008.01618.x. PMID 19126114
- [Background] Mombelli A, Decaillet F. The characteristics of biofilms in peri-implant disease. J Clin Periodontol. 2011 Mar;38 Suppl 11:203-13. doi: 10.1111/j.1600-051X.2010.01666.x. PMID 21323716
- [Background] Perez-Chaparro PJ, Duarte PM, Shibli JA, Montenegro S, Lacerda Heluy S, Figueiredo LC, Faveri M, Feres M. The Current Weight of Evidence of the Microbiologic Profile Associated With Peri-Implantitis: A Systematic Review. J Periodontol. 2016 Nov;87(11):1295-1304. doi: 10.1902/jop.2016.160184. Epub 2016 Jul 15. PMID 27420109
- [Background] Persson GR, Renvert S. Cluster of bacteria associated with peri-implantitis. Clin Implant Dent Relat Res. 2014 Dec;16(6):783-93. doi: 10.1111/cid.12052. Epub 2013 Mar 25. PMID 23527870
- [Background] Pommer B, Haas R, Mailath-Pokorny G, Furhauser R, Watzek G, Busenlechner D, Muller-Kern M, Kloodt C. Periimplantitis Treatment: Long-Term Comparison of Laser Decontamination and Implantoplasty Surgery. Implant Dent. 2016 Oct;25(5):646-9. doi: 10.1097/ID.0000000000000461. PMID 27504533
- [Background] Renvert S, Polyzois I. Treatment of pathologic peri-implant pockets. Periodontol 2000. 2018 Feb;76(1):180-190. doi: 10.1111/prd.12149. Epub 2017 Nov 29. PMID 29239086
- [Background] Romeo E, Ghisolfi M, Murgolo N, Chiapasco M, Lops D, Vogel G. Therapy of peri-implantitis with resective surgery. A 3-year clinical trial on rough screw-shaped oral implants. Part I: clinical outcome. Clin Oral Implants Res. 2005 Feb;16(1):9-18. doi: 10.1111/j.1600-0501.2004.01084.x. PMID 15642026
- [Background] Romeo E, Lops D, Chiapasco M, Ghisolfi M, Vogel G. Therapy of peri-implantitis with resective surgery. A 3-year clinical trial on rough screw-shaped oral implants. Part II: radiographic outcome. Clin Oral Implants Res. 2007 Apr;18(2):179-87. doi: 10.1111/j.1600-0501.2006.01318.x. PMID 17348882
- [Background] Schmalz G, Tsigaras S, Rinke S, Kottmann T, Haak R, Ziebolz D. Detection of five potentially periodontal pathogenic bacteria in peri-implant disease: A comparison of PCR and real-time PCR. Diagn Microbiol Infect Dis. 2016 Jul;85(3):289-294. doi: 10.1016/j.diagmicrobio.2016.04.003. Epub 2016 Apr 9. PMID 27142589
- [Background] Schwarz F, Derks J, Monje A, Wang HL. Peri-implantitis. J Periodontol. 2018 Jun;89 Suppl 1:S267-S290. doi: 10.1002/JPER.16-0350. PMID 29926957
- [Background] Toma S, Brecx MC, Lasserre JF. Clinical Evaluation of Three Surgical Modalities in the Treatment of Peri-Implantitis: A Randomized Controlled Clinical Trial. J Clin Med. 2019 Jul 3;8(7):966. doi: 10.3390/jcm8070966. PMID 31277265
- [Background] Zheng H, Xu L, Wang Z, Li L, Zhang J, Zhang Q, Chen T, Lin J, Chen F. Subgingival microbiome in patients with healthy and ailing dental implants. Sci Rep. 2015 Jun 16;5:10948. doi: 10.1038/srep10948. PMID 26077225
- [Background] Zhuang LF, Watt RM, Mattheos N, Si MS, Lai HC, Lang NP. Periodontal and peri-implant microbiota in patients with healthy and inflamed periodontal and peri-implant tissues. Clin Oral Implants Res. 2016 Jan;27(1):13-21. doi: 10.1111/clr.12508. Epub 2014 Nov 14. PMID 25399962
- [Background] Stavropoulos A, Bertl K, Eren S, Gotfredsen K. Mechanical and biological complications after implantoplasty-A systematic review. Clin Oral Implants Res. 2019 Sep;30(9):833-848. doi: 10.1111/clr.13499. Epub 2019 Jul 17. PMID 31254417
- [Background] Keeve PL, Koo KT, Ramanauskaite A, Romanos G, Schwarz F, Sculean A, Khoury F. Surgical Treatment of Periimplantitis With Non-Augmentative Techniques. Implant Dent. 2019 Apr;28(2):177-186. doi: 10.1097/ID.0000000000000838. PMID 30475243
- [Background] Serino G, Turri A. Outcome of surgical treatment of peri-implantitis: results from a 2-year prospective clinical study in humans. Clin Oral Implants Res. 2011 Nov;22(11):1214-20. doi: 10.1111/j.1600-0501.2010.02098.x. Epub 2011 Feb 11. PMID 21309860
- [Background] Carcuac O, Derks J, Abrahamsson I, Wennstrom JL, Petzold M, Berglundh T. Surgical treatment of peri-implantitis: 3-year results from a randomized controlled clinical trial. J Clin Periodontol. 2017 Dec;44(12):1294-1303. doi: 10.1111/jcpe.12813. Epub 2017 Nov 10. PMID 28902426
- [Background] Figuero E, Graziani F, Sanz I, Herrera D, Sanz M. Management of peri-implant mucositis and peri-implantitis. Periodontol 2000. 2014 Oct;66(1):255-73. doi: 10.1111/prd.12049. PMID 25123773
- [Background] Renvert S, Persson GR, Pirih FQ, Camargo PM. Peri-implant health, peri-implant mucositis, and peri-implantitis: Case definitions and diagnostic considerations. J Periodontol. 2018 Jun;89 Suppl 1:S304-S312. doi: 10.1002/JPER.17-0588. PMID 29926953
- [Background] Fu JH, Wang HL. Breaking the wave of peri-implantitis. Periodontol 2000. 2020 Oct;84(1):145-160. doi: 10.1111/prd.12335. PMID 32844418
- [Background] Roccuzzo A, Stahli A, Monje A, Sculean A, Salvi GE. Peri-Implantitis: A Clinical Update on Prevalence and Surgical Treatment Outcomes. J Clin Med. 2021 Mar 6;10(5):1107. doi: 10.3390/jcm10051107. PMID 33800894
- [Background] Schwarz F, Jepsen S, Obreja K, Galarraga-Vinueza ME, Ramanauskaite A. Surgical therapy of peri-implantitis. Periodontol 2000. 2022 Feb;88(1):145-181. doi: 10.1111/prd.12417. PMID 35103328
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Background] Schwarz F, Ferrari D, Popovski K, Hartig B, Becker J. Influence of different air-abrasive powders on cell viability at biologically contaminated titanium dental implants surfaces. J Biomed Mater Res B Appl Biomater. 2009 Jan;88(1):83-91. doi: 10.1002/jbm.b.31154. PMID 18615487
- [Background] Tastepe CS, van Waas R, Liu Y, Wismeijer D. Air powder abrasive treatment as an implant surface cleaning method: a literature review. Int J Oral Maxillofac Implants. 2012 Nov-Dec;27(6):1461-73. PMID 23189298
- [Background] Meyle J. Mechanical, chemical and laser treatments of the implant surface in the presence of marginal bone loss around implants. Eur J Oral Implantol. 2012;5 Suppl:S71-81. PMID 22834396
- [Background] Faggion CM Jr, Listl S, Fruhauf N, Chang HJ, Tu YK. A systematic review and Bayesian network meta-analysis of randomized clinical trials on non-surgical treatments for peri-implantitis. J Clin Periodontol. 2014 Oct;41(10):1015-25. doi: 10.1111/jcpe.12292. Epub 2014 Aug 11. PMID 25039292
- [Background] Blanco C, Pico A, Dopico J, Gandara P, Blanco J, Linares A. Adjunctive benefits of systemic metronidazole on non-surgical treatment of peri-implantitis. A randomized placebo-controlled clinical trial. J Clin Periodontol. 2022 Jan;49(1):15-27. doi: 10.1111/jcpe.13564. Epub 2021 Oct 28. PMID 34713471